CLINICAL TRIAL: NCT03630874
Title: Evaluation of a Prescription Support-tool for Chronic Management of Oral Antithrombotic Combinations in Adults: Protocol of a Randomized Controlled Trial Using Clinical Vignettes
Brief Title: A Prescription Support Tool for Oral Antithrombotic Combinations
Acronym: COMBI-AT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Sorbonne University (Other); Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 18-492
Record Dates: First submitted 2018-07-09; First posted 2018-08-15 (Actual); Last update posted 2019-05-16 (Actual); Status verified 2018-07

CONDITIONS: Antithrombotics Prescriptions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental arm (Experimental)
  Interventions: Other: Evaluate the impact of a prescription support tool
- Control arm (No Intervention): Selected physicians will receive 3 different clinical vignettes, each corresponding to a specific situation for which the physician will have to indicate (without the tool) the "right prescription" of ATs by answering a multiplechoice question, with the number, type, duration and dosage of AT provided.

INTERVENTIONS:
Other: Evaluate the impact of a prescription support tool — From a systematic review of international guidelines (2012-2018), we developed a prescription support-tool synthesizing national and international guidelines on chronic management (≥ 1 month) of oral AT agents without considering in-hospital management and bridging therapy.
  In the experimental group, the tool will be provided with an explanatory guide. Selected physicians will receive 3 different clinical vignettes, each corresponding to a specific situation for which the physician will have to indicate (thanks to the tool) the "right prescription" of ATs by answering a multiple-choice question, with the number, type, duration and dosage of AT provided.
  Arms: Experimental arm

SUMMARY:
From a systematic review of international guidelines (2012-2018), a prescription support-tool synthesizing national and international guidelines on chronic management (≥ 1 month) of oral AT agents without considering in-hospital management and bridging therapy will be developed. Guidelines dealing with the use of oral ATs for non-valvular atrial fibrillation, coronary artery disease, ischemic stroke, valvular heart disease, peripheral artery disease and venous thromboembolism in adults will be included. These pathologies were selected because most prescriptions of ATs are related to neuro-cardiovascular diseases and because this study would provide a synthesis relevant for clinicians in charge of the follow-up of patients with oral AT combinations. Studies are needed to assess the impact of this tool on appropriate prescribing.

DETAILED DESCRIPTION:
Oral antithrombotic (AT) drugs are widely implicated in serious and preventable bleeding events, which justifies the implementation of risk minimization actions. Avoiding inappropriate oral AT combinations is a major concern, particularly for patients with multiple chronic conditions. The first step is to provide fast and easy access to the latest recommendations. From a systematic review of international guidelines (2012-2018), a prescription support-tool synthesizing national and international guidelines on chronic management (≥ 1 month) of oral AT agents without considering in-hospital management and bridging therapy will be developed. Our main objective in this study is to evaluate the accuracy of this tool by measuring the appropriateness of oral AT prescriptions according to the most recent guidelines.

Methods and analysis: In this web-based randomized controlled trial, participating French general practitioners and cardiologists in the outpatient setting will be randomized by use or not of the prescription support-tool. They will be asked to provide the number of drugs, drug class, duration and dosage of ATs, within a time window of 10 minutes, for 3 different clinical situations presented as clinical vignettes (multiple-choice questions). The scientific committee has created and validated 30 clinical vignettes illustrating outpatient clinical situations for which the use of oral ATs (single, dual or triple therapy) is recommended or not according to the guidelines. All data will be treated anonymously.

Ethics and dissemination: If the prescription support-tool is associated with more appropriate prescription of AT combinations, its dissemination to further evaluate outcome data including haemorrhage, ischemic events, and death will be considered.

ELIGIBILITY:
Inclusion Criteria:

* French practicing physicians who are involved in outpatient settings, including general practitioners and cardiologists.

Exclusion Criteria:

* Physicians with an exclusive hospital practice.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 478 (Actual)
Dates: Start 2018-11-05 (Actual); Primary Completion 2019-02-14 (Actual); Study Completion 2019-02-14 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure is the rate of the "right prescription of oral ATs" as defined according to the guidelines in terms of number, class, duration and dosage between the two groups. | Day one
  How will be defined the "right prescription of oral ATs" :
  From a systematic review of international guidelines (2012-2018), has been developed, a prescription support-tool synthesizing 70 national and international guidelines on chronic management (≥ 1 month) of oral AT agents without considering in-hospital management and bridging therapy.
  The scientific committee of this study (cardiologist, internist-geriatricians, general practitioner and epidemiologists) created and validated 30 clinical vignettes.
  The expert committee of this study had to review all clinical vignettes with the prescription support-tool (external validation) to confirm their agreement with clinical practice and their readability.
  Thus, the "right prescription of oral ATs" was defined a priori (right or false) thanks to the prescription support tool and validated by the expert committee and the scientific committee.

SECONDARY OUTCOMES:
The rate of the "right prescription of oral ATs" performed by physicians' specialty. | Day one
  Physicians' specialty: french physicians who are involved in outpatient settings, including general practitioners and cardiologists. Physicians with an exclusive hospital practice will not be considered.
The difference between the control and intervention groups in the degree of confidence physicians have in their AT prescriptions in line with the guidelines. | Day one
  The degree of confidence was defined a priori with this question: "On a scale of 0 to 10, what is your degree of confidence in the adequacy of your prescription in relation to the guidelines?"

CONTACTS AND LOCATIONS:
Overall Officials: Lorène ZERAH, M.D, Principal Investigator — APHP / INSERM

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zerah L, Bonnet-Zamponi D, Frappe P, Hauguel-Moreau M, De Rycke Y, Magnier AM, Pautas E, Charles P, Collet JP, Dechartres A, Tubach F. Evaluation of a prescription support-tool for chronic management of oral antithrombotic combinations in adults using clinical vignettes: protocol of a randomised controlled trial. BMJ Open. 2019 Jun 9;9(6):e025544. doi: 10.1136/bmjopen-2018-025544. PMID 31182442